CLINICAL TRIAL: NCT02475889
Title: Hepatic Radiofrequency Ablation Increases T Cell Infiltraion and PD-L1 Expression in Primary Tumor in Patients With Synchronous Colorectal Cancer Liver Metastases
Brief Title: Hepatic RFA Increases T Cell Infiltraion and PD-L1 Expression in Primary Colorecatl Cancer
Status: Completed | Type: Observational
Sponsor: The First People's Hospital of Changzhou (Other)
Responsible Party: Principal Investigator, Liangrong Shi, Director, The First People's Hospital of Changzhou
Other Study IDs: RFAOO2
Record Dates: First submitted 2015-06-06; First posted 2015-06-19 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Paraffin-embedded tissues of endoscopic biopsy specimen and matched resected primary tumor specimen
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- RFA group: patients who received hepatic RFA followed by primary tumor resection were assigned to the RFA group
  Interventions: Procedure: Hepatic RFA; Procedure: Primary tumor resection
- Non-RFA group: patients who received initial primary tumor resection without RFA
  Interventions: Procedure: Primary tumor resection

INTERVENTIONS:
Procedure: Hepatic RFA — Hepatic RFA was performed under guidace of ultrasonography (US) or computed tomography (CT) before primary tumor resection.
  Groups: RFA group
Procedure: Primary tumor resection — Primary tumor resection were performed pre- or post-RFA for liver metastases.

SUMMARY:
It has been shown that RFA induced systemic tumor antigen-specific T cell responses in human carcinoma. However, there are insufficient studies on the immune modulation of tumor microenviroment (TME) outside of the ablation zone. In order to study how RFA modifies TME in human cancer patients, investigators performed a retrospective study of a unique cohort of patients who suffered from synchronous CRCLM.

DETAILED DESCRIPTION:
Radiofrequency ablation (RFA) is widely used as a local treatment for tumors such as small hepatocellular carcinomas, renal cancer and solitary colorectal cancer liver metastases (CRCLM). RFA induces localized coagulation necrosis and leads to the release of large amounts of cellular debris in situ, which can serve as a source of tumor antigens to elicit host adaptive immune responses against tumors. Several studies on preclinical animal models have shown that localized tumor ablation by RFA can induce systemic T-cell mediated antitumor immunity. Antigen-specific T cell immune responses were also observed in patients with hepatic tumors after RFA therapy. However, the RFA-induced immune responses are not sufficient to prevent tumor recurrence. The underlying mechanisms remain obscure.

Programmed death-ligand 1 (PD-L1), an important immune checkpoint molecule, is often up-regulated on tumor cells and tumor associated myeloid cells. It impairs T cell-mediated immune responses upon engagement with its cognate co-inhibitory receptor PD-1, which is always highly expressed on tumor-infiltrating lymphocytes. PD-L1 expression can be induced by pro-inflammatory cytokines, especially type I interferon (IFN), as an important self-limiting mechanism to prevent rampant autoimmunity. Recent studies show that PD-L1 expression on tumor cells is associated with T cell infiltration, suggesting PD-L1 is actively involved in suppressing antitumor immune responses in the tumor microenvironment (TME). Whether the PD-L1/PD1 axis is involved in modulating the antitumor T cell immune responses induced by RFA is unclear.

The objective of this investigation was to study the RFA-induced immune responses in tumor tissues from cancer patients.

ELIGIBILITY:
Inclusion Criteria:

Patients with histologically confirmed asynchronous liver metastases received initial hepatic RFA or initial primary tumor resection.

Exclusion Criteria:

1. Preoperative CT, RT and other antitumor treatment
2. Emergency surgery
3. Initial hepatectomy
4. No qualified endoscopic biopsy

Ages: 32 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 391 consecutive patients with synchronous colorectal cancer liver metastases were initially included in this study. Among of them, 38 patients who received initial hepatic RFA followed by primary tumor resection were identified as RFA group, and the other 40 patients who received initial primary tumor resection were identified as Non-RFA group.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2007-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Number of T cell infiltraion in primary tumor | 2 weeks
  Number of T cell infiltraion in primary tumor was evaluated by immunohistochemical staining
PD-L1 expression in primary tumor | 2 weeks
  PD-L1 expression in primary tumor was evaluated by immunohistochemical staining

CONTACTS AND LOCATIONS:
Overall Officials: Changping Wu, M.D., Study Chair — The First People's Hospital of Changzhou